CLINICAL TRIAL: NCT07198971
Title: Feasibility Study Incorporating Music Therapy to Optimise the Smoking Cessation Process Coordinated by a Tobacco Addiction Nurse in Smoking Patients Being Treated for Cancer
Acronym: TEMPOS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PROICM 2025-02 TEM
Record Dates: First submitted 2025-09-09; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Cancer (With or Without Metastasis)
Keywords: Smoking cessation; music therapy; tobacco addiction treatment
MeSH Terms: conditions — Neoplasms; Smoking Cessation | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Music therapy is offered to provide additional support in the process of quitting smoking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EXPERIMENTAL (Experimental): Tabacco nurse consultation with music therapy session will be done at day 1 day 7 day 15 day 30 month 2 month 3 and month 6 (end of study)
  Interventions: Other: Music therapy

INTERVENTIONS:
Other: Music therapy — Music therapy sessions in addition to nursing consultations:
  creation of a soundtrack to listen to in order to help quit smoking

SUMMARY:
The innovative nature of this project lies in the combination of three types of intervention: tobacco addiction treatment, music therapy and therapeutic education.

Three disciplines that work together.

1. Tobacco addiction treatment: reducing consumption, quitting,
2. Music therapy: acting on emotions and reward circuits,
3. Therapeutic education: promoting independent healthy practices. Patients learn to use the soundtrack independently to help them manage withdrawal symptoms caused by reducing or stopping tobacco consumption.

In this programme, patients play an active role on several levels:

* working with the music therapist to create a personalised 'soundtrack';
* identifying situations in which music can help them manage withdrawal symptoms;
* using music independently in their everyday lives. The music therapy protocol will be proposed in this study, the soundtrack is co-created by the music therapist and the patient based on the patient's musical tastes and needs. The fact that the patient can use the musical tool independently also gives them significant leverage in their withdrawal process, allowing them to act on withdrawal symptoms and the main factors contributing to relapse.

DETAILED DESCRIPTION:
Music therapy could address the three elements mentioned above:

* add a practitioner other than the tobacco specialist,
* increase the patient's perception of self-efficacy,
* provide the patient with a personalised soundtrack that may have an effect on withdrawal symptoms associated with smoking cessation.

Music therapy could increase the chances of successful cessation. It therefore seems innovative to offer an educational intervention combining the tobacco specialist nurse and the music therapist, which would enable patients to use a musical tool co-developed with the music therapist independently at home. There are no data on the learning and use of such a tool to reinforce self-efficacy in managing smoking cessation. The analysis of the existing literature is poor in terms of music therapy and addiction and virtually non-existent in terms of tobacco addiction.

The objective is to evaluate the feasibility of an intervention combining tobacco addiction treatment and music therapy and its impact on smoking cessation symptoms in patients with cancer who smoke.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over the age of 18
2. Patients with tobacco-related or non-tobacco-related cancer (excluding blood cancer)
3. Patients who smoke daily
4. Patients wishing to begin a smoking cessation programme
5. Patients with a prognosis of > 1 year
6. Patients who have given their informed, written and express consent
7. Patients affiliated with a French social security scheme

Exclusion Criteria:

1. Patients with uncorrected hearing loss
2. Patients with unstable psychiatric conditions
3. Patients for whom regular follow-up is impossible for psychological, family, social or geographical reasons
4. Patients under guardianship, curatorship or judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who adhered to the supervised sessions, combining follow-up by a tobacco addiction nurse and follow-up in music therapy | From baseline to month 6
  The patient is considered compliant if they have participated in 4 or more of the 6 supervised sessions combining tobacco addiction consultations

SECONDARY OUTCOMES:
Tobacco use | at baseline, at month 3, at month 6
  Number of cigarettes smoked per day and Measurement of exhaled CO and Tobacco dependence scale score: Simplified Fagerström Test
Withdrawal symptoms | at baseline, at month 3, at month 6
  Scores on the Smoking Cessation Scale
The craving | at baseline, at month 3, at month 6
  Scores obtained on the French Tobacco Craving Questionnaire
Motivation | at baseline, at month3, at month 6
  Scores on the 0-10 Digital Scale assessing motivation
Confidence | at baseline, at month 3, at month 6
  Scores on the EN assessing confidence
Sense of personal competence | at baseline, at month 3, at month 6
  General Self Efficacy Scale questionnaire
Symptoms of anxiety and depression | at baseline, at month 3, at month 6
  Anxiety and depression scores on the Hospital Anxiety and Depression Scale
Describe adherence to independent listening in music therapy between T2 and T6. | at baseline, at month 3 and at month 6
  Describe the number of times the patient listened to the audio recording per day, as recorded in a logbook.

CONTACTS AND LOCATIONS:
Overall Officials: GONZALEZ Marie Laure, Tobacco Nurse, Principal Investigator — marie-laure.gonzalez@icm.unicancer.fr
Locations (1):
- Institut Du Cancer de Montpellier, Montpellier, Herault, France

IPD SHARING:
Plan to Share IPD: No
Participant data will be made available on request and with completion of a contract between the sponsor and the requester

REFERENCES:
- [Background] Benowitz NL. Neurobiology of nicotine addiction: implications for smoking cessation treatment. Am J Med. 2008 Apr;121(4 Suppl 1):S3-10. doi: 10.1016/j.amjmed.2008.01.015. PMID 18342164
- [Background] Jassem J. Tobacco smoking after diagnosis of cancer: clinical aspects. Transl Lung Cancer Res. 2019 May;8(Suppl 1):S50-S58. doi: 10.21037/tlcr.2019.04.01. PMID 31211105
- [Background] Kathuria H, Neptune E. Primary and Secondary Prevention of Lung Cancer: Tobacco Treatment. Clin Chest Med. 2020 Mar;41(1):39-51. doi: 10.1016/j.ccm.2019.10.002. PMID 32008628
- [Background] Tabac. (https://www.who.int/fr/news-room/fact-sheets/detail/tobacco). Accessed 7 December 2023.
- [Background] Tabac - Réduire les risques de cancer. (https://www.e-cancer.fr/Comprendre-prevenir-depister/Reduire-les-risques-de-cancer/Tabac). Accessed 15 December 2023.